CLINICAL TRIAL: NCT07024966
Title: Effect of the Combination of Pterostilbene Cocrystal With Silybin and Nicotinamide Riboside on High-Intensity Exercise-Induced Oxidative Stress: A Randomized, Crossover, Placebo-Controlled, Triple-Blind Study
Brief Title: Effect of the Combination of Pterostilbene Cocrystal With Silybin and Nicotinamide Riboside on Exercise-Induced Oxidative Stress
Acronym: PT-SILAOX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Eurecat (Other)
Collaborators: Circe, S.L. (Unknown)
Responsible Party: Principal Investigator, Antoni Caimari, Director of the of the Biotechnology Area, Fundació Eurecat
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PT-SILAOX
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Oxidative Stress; Physical Activity; Antioxidant Effect
Keywords: Oxidative Stress; High-intensity exercise; Pterostilbene; Antioxidant supplement; Nutraceutical; Crossover trial; Exercise recovery; Nutritional intervention; Polyphenols; Cocrystal
MeSH Terms: conditions — Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants treated with Microcrystalline Cellulose for 14 days
  Interventions: Dietary Supplement: Control Group
- ccPT-SIL-NR Group (Experimental): Participants treated with pterostilbene, silybin, and nicotinamide riboside for 14 days
  Interventions: Dietary Supplement: Pterostilbene-silybin-nicotinamide riboside

INTERVENTIONS:
Dietary Supplement: Pterostilbene-silybin-nicotinamide riboside — Participants will take 2 sachets, each containing 340 mg of ccPT, silybin and nicotinamide riboside, and 1.91 g of excipients.
  Arms: ccPT-SIL-NR Group
Dietary Supplement: Control Group — Participants will take 2 sachets, each containing 340 mg microcrystalline cellulose, and 1.91 g of excipients.
  Arms: Placebo

SUMMARY:
This study aims to evaluate the effects of the dietary supplement ccPT-SIL-NR, which contains pterostilbene (ccPT), silybin (SIL), and nicotinamide riboside (NR), on oxidative stress markers after a high-intensity exercise session. The primary objective is to assess changes in blood malondialdehyde (MDA) levels.

Secondary objectives include evaluating the effects on oxidative DNA damage (8-OHdG), lipid peroxidation (F2-isoprostanes), total antioxidant capacity (FRAP assay), glutathione ratio (GSH/GSSG), antioxidant enzyme activity (SOD, CAT, GPx), inflammatory markers (hsCRP, MCP-1, IL-6), muscle damage markers (LDH, CK), cortisol levels, renal function (creatinine), and gene expression patterns through transcriptomic analysis.

The study will include 14 healthy male participants in a randomized, tripple-blind, placebo-controlled, crossover design. Each participant will receive both the ccPT-SIL-NR supplement and placebo for 14 days each, separated by a washout period of at least one week. A high-intensity exercise test will be performed at the end of each supplementation period. Total study duration per participant will be a minimum of 6 weeks.

DETAILED DESCRIPTION:
This study aims to evaluate the effect of a nutritional supplement combining pterostilbene, silybin, and nicotinamide riboside on oxidative stress induced by high-intensity exercise. Oxidative stress occurs when there is an imbalance between the production of reactive oxygen species and the body's ability to counteract their harmful effects. High-intensity physical activity is known to increase oxidative stress, potentially leading to cellular damage and inflammation. The supplement under investigation has shown antioxidant properties in preclinical models, and this trial seeks to explore its efficacy in humans. The trial is a randomized, triple-blind, placebo-controlled, and crossover study. Fourteen healthy, physically active men aged 18-50 will be recruited. Each participant will take either the supplement or placebo twice daily for 14 days, followed by a treadmill exercise session at 80% of their VO₂ max. After a washout period, participants will switch treatments and repeat the protocol. Blood and urine samples will be collected both at baseline (prior to supplement intake and without any physical activity) and after the exercise test to evaluate markers of oxidative stress, inflammation, muscle damage, and antioxidant capacity. The main outcome is the change in plasma levels of malondialdehyde (MDA). Secondary outcomes include urinary 8-OHdG and F2-isoprostanes, antioxidant enzyme activities, cortisol levels, and gene expression profiles. This study will help to determine whether the supplement can mitigate exercise-induced oxidative stress and support recovery in recreational athletes.

Participants will attend seven in-person visits:

* V0; week 0 (Screening): Informed consent, eligibility check, medical history, anthropometry.
* V1; week 1 (Baseline 1): Pre-intervention samples collection, supplement/placebo dispensation.
* V2; week 1: Exercise test to determine VO₂ max.
* V3; week 3: First treadmill session after 14 days of intervention with the supplement or placebo, blood draw.
* V4; week 3: Urine sample drop-off post-exercise (0-3h and 3-24h).
* V5; week 4 (Baseline 2): Pre-second intervention samples, crossover begins.
* V6; week 6: Second treadmill session, blood draw.
* V7; week 6: Final urine collection post-exercise (0-3h and 3-24h)..

ELIGIBILITY:
Inclusion Criteria:

* Male participants between 18 and 50 years of age who are amateur runners.
* Engage in at least 3 continuous running sessions per week, each lasting 60 minutes, which corresponds to a high level of physical activity according to the International Physical Activity Questionnaire (IPAQ).*
* Self-report being able to continuously run for 45 minutes at high intensity without difficulty.
* Provide signed informed consent prior to participation in the study.
* Able to read, write, and speak either Catalan or Spanish.

  * High level of physical activity according to the IPAQ: vigorous physical activity (such as running) on at least 3 days per week, with a total energy expenditure ≥1500 MET-min/week.

MET value for vigorous activity = 8 × minutes × days per week.

Exclusion Criteria:

* Body Mass Index (BMI) ≤ 18 kg/m² or ≥ 30 kg/m².
* Presence of chronic diseases associated with increased oxidative stress, such as diabetes, hypertension, chronic obstructive pulmonary disease (COPD), or neurodegenerative diseases.
* Personal history of cardiovascular disease, including myocardial infarction, angina pectoris, stroke, or peripheral artery disease.
* Use of antibiotics within 30 days prior to study entry.
* Use of medications or vitamin supplements that may interfere with the study supplement and exceed 100% of the recommended daily intake within 30 days prior to the start of the study.
* Use of polyphenol supplements, herbal extracts, or phytotherapeutic products that may interfere with the study treatment within 30 days prior to study start.
* Alcohol consumption of 4 or more Standard Drink Units (SDUs) per day or 28 SDUs per week.*

  *One SDU is defined as 10 grams of alcohol. This corresponds approximately to: 1 glass of wine (120 mL), 1 beer (330 mL), or 1 small spirit (25 mL); 2 SDUs correspond to 1 glass of brandy or liqueur (55 mL), 1 whiskey (70 mL), or a mixed drink (75 mL).
* Active smoker.
* Unintentional weight loss of more than 3 kg in the past 3 months.
* Known food allergies and/or intolerances related to the study products.
* Presence of anemia.
* Presence of chronic gastrointestinal diseases* or cancer.**

  *Chronic gastrointestinal diseases include those in an active phase that may interfere with nutrient absorption. Common examples include gastritis, hiatal hernia, Crohn's disease, celiac disease, irritable bowel syndrome, diverticulitis, diverticulosis, chronic constipation, and ulcerative colitis.

  **Individuals with a history of cancer may be included only if they are in complete remission at the start of the study.
* Participation in another drug clinical trial or nutritional intervention study within 30 days prior to study inclusion.
* Inability to follow the study guidelines.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Malondialdehyde (MDA) plasma levels | At week 1, week 3, week 4 and week 6.
  Plasma MDA levels will be measured using commercial ELISA kits

SECONDARY OUTCOMES:
Age | At week 0 (pre-selection visit)
  The age of the volunteers will be recorded in the case report form.
Height (cm) | At week 0 (pre-selection visit)
  Height measured with standardized method
Body Weight (Kg) | At week 0 (pre-selection visit)
  Weight measured using the InBody 970 device
Body Mass Index (BMI) (Kg/m^2) | At week0 (pre-selection visit)
  Weight and height will be combined to report BMI in kg/m^2
Urine 8-hydroxy-2'-deoxyguanosine (8-OHdG) levels | At week 1, week 3, week 4 and week 6.
  Urine 8-OHdG levels will be measured using commercial ELISA kits
Urine F2-isoprostanes levels | At week 1, week 3, week 4 and week 6.
  Urine F2-isoprostanes levels will be measured using commercial ELISA kits
Plasma antioxidant capacity | At week 1, week 3, week 4 and week 6.
  Plasma antioxidant capacity will be measured by the Ferric Reducing Antioxidant Power assay using ELISA kits.
Erythrocyte Redox Status (GSH/GSSG Ratio) | At week 1, week 3, week 4 and week 6.
  The ratio of reduced glutathione (GSH) to oxidized glutathione (GSSG) will be measured in erythrocytes using commercial ELISA kits.
Superoxide Dismutase (SOD) Activity | At week 1, week 3, week 4 and week 6.
  Serum levels of superoxide dismutase (SOD) activity will be measured using a commercial ELISA kit.
Catalase (CAT) Activity | At week 1, week 3, week 4 and week 6.
  Serum catalase (CAT) activity will be measured using a commercial ELISA kit.
Glutathione Peroxidase (GPx) Activity | At week 1, week 3, week 4 and week 6.
  Serum levels of glutathione peroxidase (GPx) activity will be measured using a commercial ELISA kit.
Serum High-Sensitivity C-Reactive Protein (hs-CRP) Levels | At week 1, week 3, week 4 and week 6.
  Serum levels of high-sensitivity C-reactive protein (hs-CRP) will be measured using turbidimetric methods.
Plasma Monocyte Chemoattractant Protein-1 (MCP-1) Levels | At week 1, week 3, week 4 and week 6.
  Plasma levels of monocyte chemoattractant protein-1 (MCP-1) will be measured using a commercial multiplex Cytometric Bead Array kit.
Plasma Interleukin-6 (IL-6) Levels | At week 1, week 3, week 4 and week 6.
  Plasma levels of interleukin-6 (IL-6) will be measured using a commercial multiplex Cytometric Bead Array kit.
Plasma Lactate Dehydrogenase (LDH) Levels | At week 1, week 3, week 4 and week 6.
  Plasma levels of lactate dehydrogenase (LDH) will be measured using commercial ELISA kits.
Plasma Creatine Kinase (CK) Levels | At week 1, week 3, week 4 and week 6.
  Plasma levels of creatine kinase (CK) will be measured using commercial ELISA kits
Serum Cortisol Levels | At week 1, week 3, week 4 and week 6.
  Serum cortisol levels will be determined using electrochemiluminescence methods.
Urinary Creatinine Levels | At week 1, week 3, week 4 and week 6.
  Urinary creatinine levels will be measured using a commercial ELISA kit
Maximal Oxygen Uptake (VO₂ max) | At week 1.
  VO₂ max. be assessed through a graded exercise test. This data will be used to calibrate subsequent treadmill sessions at 80% of each participant's VO₂ max.
Heart Rate, Treadmill Speed and Incline | At week 1.
  Heart rate, treadmill speed, and incline at the intensity of 80% of each participant's VO₂ max. will be recorded in the case report form.
Physical Activity Level (Questionnaire-Based) | At week 0, week 1, week 3, week 4 and week 6.
  Physical activity level will be assessed using the "Quick Physical Activity Classifier" questionnaire, adapted from the PEFS Guide of the Catalan Government.
Whole Blood Transcriptomic Profile (RNA-seq) | At week 1, week 3, week 4 and week 6.
  Gene expression will be analyzed in whole blood samples preserved in PAXgene Blood RNA tubes.
Concomitant medication | At week 0, week 1, week 3, week 4 and week 6.
  The use of any concomitant medication will be recorded through participant-reported entries in the case report form.
Heart Rate | At week 0, week 1, week 3, week 4 and week 6.
  Heart rate will be measured using the Omron HEM-907 monitor.
Systolic Blood Pressure | At week 0, week 1, week 3, week 4 and week 6.
  Systolic Blood Pressure will be measured using the Omron HEM-907 monitor.
Diastolic Blood Pressure | At week 0, week 1, week 3, week 4 and week6.
  Diastolic Blood Pressure will be measured using the Omron HEM-907 monitor.
Use of Dietary Supplements | At week 0, week 1, week 3, week 4 and week 6.
  Dietary supplements consumed during the study will be recorded in the case report form.
Intervention Compliance (Supplement Intake Adherence) | At week 3 and week 6.
  Compliance with the intervention will be assessed indirectly by calculating the ratio between the number of supplement sachets theoretically assigned and the number actually consumed.
Adverse events | At week 3 and week 6.
  Possible adverse events derived from taking study's products will be recorded in the case report form

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Caimari, PhD, Principal Investigator — Fundació Eurecat
Locations (1):
- Fundació Eurecat, Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Technological Centre of Nutrition and Health. Eurecat_Reus. — http://eurecat.org